CLINICAL TRIAL: NCT07211282
Title: Transmural Physical Activity Monitoring and Guidance During Phase 3 Cardiac Rehabilitation: the Antwerp Activity Index
Brief Title: Monitoring and Guidance of Physical Activity During the Maintenance Phase of Cardiac Rehabilitation: the Antwerp Activity Index
Acronym: AMAAI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BUN3002025000061; G084023N (Other Grant/Funding Number: Fonds Wetenschappelijk Onderzoek (FWO))
Record Dates: First submitted 2025-09-04; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Rehabilitation; Cardiovascular Disease Prevention
Keywords: physical activity; cardiac rehabilitation; heart rate monitor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AAI usage through personalised target (Experimental): Participants are instructed to continuously wear a Fitbit Versa 4 smartwatch for the whole monitoring period, sync the data daily via the Fitbit application, and charge the device when needed. The intervention group has access to the generated AAI scores through a study application. During an initiation visit, they will be informed about how the score works and its purpose. They will receive tailored targets to adhere to. This group will also receive semi-automatic feedback reports through the study application. Feedback will be provided every two weeks for the first two months and once more at the end of the third month. No feedback will be given during the last month of follow-up.
  Interventions: Device: Activity score
- Blinded AAI data collection (No Intervention): Participants are instructed to continuously wear a Fitbit Versa 4 smartwatch for the whole monitoring period, sync the data daily via the Fitbit application, and charge the device when needed. They can use the device to their liking. They do not have access to the AAI algorithm, nor will they receive feedback through the study application.

INTERVENTIONS:
Device: Activity score — 4 month follow-up and feedback from a heart rate and personal characteristics based activity score.
  Arms: AAI usage through personalised target

SUMMARY:
The goal of this clinical trial is to determine whether the AAI activity score can help cardiac rehabilitation patients adhere to physical activity guidelines after participating in an in-hospital cardiac rehabilitation program. The main questions it aims to answer are:

1. Does the AAI activity score have an impact on adherence to physical activity maintenance during phase 3 CR?
2. Does the AAI activity score predict changes in cardiorespiratory fitness? Researchers will compare participants who use the AAI activity score with those who do not to determine if there are differences in physical activity adherence.

Participants will:

* Wear a smartwatch to continuously measure heart rate for 4 months;
* Perform an exercise stress test at the end of the study;
* Fill in several questionnaires at the end of the study.

DETAILED DESCRIPTION:
Adopting and maintaining an active lifestyle after phase 2 cardiac rehabilitation (CR) is crucial for cardiac patients. Tools to provide an active transition from phase 2 CR to phase 3 CR are lacking, resulting in negative changes in physical activity (PA) behaviour, cardiovascular risk profiles and cardiorespiratory fitness (CRF) levels. The researchers developed a procedure that calculates a PA-score (Antwerp Activity Index; AAI) based on reliable heart rate (HR) data collected by commercially available heart rate monitors (HRMs), which is designed to reflect changes in CRF. This procedure could serve as a valuable tool to facilitate a more active transition from phase 2 CR to phase 3 CR. Ultimately, positively influencing CR patients' PA levels (and possibly) cardiovascular and overall health-related outcomes.

This study will collect HR data with the Fitbit Versa 4 smartwatch and Polar H10 chest strap with the aim of:

Goal 1. Assessing the effect of our AAI-score intervention on adherence towards physical activity maintenance of post-phase 2 CR patients during phase 3 CR.

Goal 2. Assessing the potential differences in the participants' self-experienced physical activity and objectively measured physical activity.

Goal 3. Investigating the correlation between adherence to our AAI score and changes in CRF.

Goal 4. Measuring the adherence to our AAI score intervention. Goal 5. For a subpopulation of AF patients, we will analyse whether the AAI score intervention influences AF recurrence and burden.

Goal 6. Analysing technical outcomes regarding the use of the AAI score and the accompanying application. This will include system performance as well as user interaction with different elements of the application.

Patients complying with the inclusion criteria who completed phase 2 CR of two large care facilities and who are interested will be randomised into one of two groups:

Group 1: Patients who, after following the standard multidisciplinary in-hospital phase 2 CR trajectory, receive a Fitbit Versa 4 and our application with our AAI-score and who receive regular feedback (intervention group).

Group 2: Patients who, after following the standard multidisciplinary in-hospital phase 2 CR trajectory, receive a Fitbit Versa 4 with blinded AAI data collection and no feedback (control group - standard care).

Participants start with a run-in period wherein their eligibility for continuous PPG-HR tracking will be objectively measured. Objective eligibility will be determined by correlation of the Fitbit HR with the Polar HR (Polar H10 chest strap). The eligibility assessment will take place in the three consecutive CR training sessions scheduled for the participant. If deemed ineligible, the participant's participation in the study ends. Participants deemed eligible during the run-in period will be randomised to the intervention or control group.

All included participants will use the Fitbit device for an average of four months. Patients are instructed to continuously wear the Fitbit Versa 4 smartwatch for the whole monitoring period, sync the data daily via the Fitbit application, and charge the device when needed. The intervention group has access to the generated AAI scores through a study application. During an initiation visit, participants will be informed about how the score works and its purpose. The intervention group will receive tailored targets to adhere to. This group will also receive semi-automatic feedback reports through the application. Feedback will be provided every two weeks for the first two months and once more at the end of the third month. No feedback will be given during the last month of follow-up. Feedback is solely based on the collected scores and not on the values used to calculate the score (heart rate). Feedback is limited to overviews of recent days and motivational messages aimed at maintaining or increasing their scores. The control group also receives the Fitbit device but does not have access to the scores generated by the AAI algorithm or receive feedback through the Cardio2U application. This simulates current standard care. The AF subpopulation of both groups will also receive a license to use the FibriCheck application for the duration of the study. An application of the same name will accompany this. These measurements are taken in the background without participant intervention. At the end of the 4-month follow-up period, both the intervention and control groups will perform an exercise stress test. At this moment, the study ends, and all related devices are returned to a study team member. During this visit, a study team member will assist participants in completing two IPAQ questionnaires, which will assess their PA levels over the last two weeks. Through a personal online link, participants will also be asked to complete a quality of life questionnaire (SF-36), a self-developed experience questionnaire (PREM) and a digital health readiness questionnaire (DHRQ). The use of the AAI score through the application will be monitored throughout the entire study period, which occurs automatically without participant intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years,
2. Patients in the last phase of phase 2 CR,
3. Having a smartphone available,
4. Being capable of signing the informed consent.

Exclusion Criteria:

1. Patients with high-risk criteria for safe exercise participation following a cardiac event, including:

   1. Ejection fraction less than 30%
   2. Decrease in systolic blood pressure of more than 15 mmHg with exercise
   3. Serious arrhythmias at rest or exercise-induced
   4. Exercise-induced ischemia indicated by angina more than 2 mm ST segment depression on the ECG
2. Patients with severe heart failure (NYHA III-IV),
3. Patients with implantable devices (e.g. pacemakers),
4. Patients diagnosed with permanent AF,
5. Patients who do not speak and read Dutch or English,
6. Patients who have cognitive impairment (e.g. severe dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Objective moderate-to-vigorous physical activity performance adherence | From enrollment to the end of treatment at 4 months
  The primary aim of this study is to assess the impact of using the developed AAI score on adherence to moderate-to-vigorous pysical activity (MVA) during phase 3 CR. This will be objectively measured and analysed by calculating the number of minutes per week a participant spends above the threshold for moderate-to-vigorous physical activity, determined using individualised heart rate zones derived from cardiopulmonary exercise testing (CPET). Continuous heart rate data (collected using the Fitbit device) are used to calculate total MVPA minutes per week.
Subjective moderate-to-vigorous physical activity performance adherence | From enrollment to the end of treatment at 4 months
  At the end of the study, during the final study visit, researchers will question participants on their PA over the last 14 days using the International Physical Activity Questionnaire (IPAQ), a validated instrument for measuring short-term PA behaviour. The responses are used to calculate an activity level in Metabolic Equivalent of Task (MET)-minutes per week.

SECONDARY OUTCOMES:
Difference in MET-minutes/week in objectively measured physical activity and subjectively reported physical activity. | From enrollment to the end of treatment at 4 months.
  The researchers aim to analyse differences between self-reported (subjective) and objectively measured physical activity (PA) adherence, to provide a comprehensive overview of guideline adherence. For comparability, objectively measured data will be expressed in MET-minutes per week, calculated as the product of minutes spent in each intensity zone (moderate or vigorous) multiplied by the corresponding MET intensity as defined in the IPAQ scoring protocol.
Correlation between adherence to AAI score and cardiorespiratory fitness changes, as measured by VO2peak. | from entrollment to the end of treatment at 4 months.
  The researchers investigate whether adherence to the AAI score, measured as the percentage of days the target is reached, correlates with changes in CRF, measured through VO2peak.
Percentage of days participants adhere to AAI score target. | From enrollment to the end of treatment at 4 months.
  To assess whether patients adhere to the instructions and goals set by the AAI application. The percentage of days participants adhere to the daily target score will be calculated.
Activity score influence on AF burden and recurrence. | From enrollment to the end of treatment at 4 months.
  The Fibricheck application will measure the burden of AF within a specific subset of patients diagnosed with AF through semi-continuous PPG measurements. This burden will be objectified as the proportion of measurements with AF in relation to the total number of measurements taken.

OTHER OUTCOMES:
Up/down time of the activity score system and application. | From enrollment to the end of treatment at 4 months.
  System availability will be quantified as the proportion of time the application and algorithm were operational during the study period. Uptime percentage will be calculated as the total hours the system was available divided by the total hours in the observation period) × 100. Downtime will be reported as the cumulative duration (in hours or days) the system was not usable, expressed both in absolute terms and as a percentage of the total study period.

CONTACTS AND LOCATIONS:
Overall Officials: Hein Heidbuchel, Principal Investigator — University Hospital, Antwerp
Locations (2):
- Belgium (2):
  - University Hospital Antwerp, Edegem, Antwerp
  - Jessa Hospital Hasselt, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No
Study data will be presented on a group rather than individual participant level.